CLINICAL TRIAL: NCT00073112
Title: A Phase 2 Study of ABT-751 in Subjects With Refractory Colorectal Carcinoma
Brief Title: A Study of ABT-751 in Patients With Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-416; NCT00080717 (obsolete NCT alias)
Record Dates: First submitted 2003-11-17; First posted 2003-11-18 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — ABT751

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ABT-751

SUMMARY:
The purpose of the study is to determine if ABT-751 will decrease tumors, and determine how long the tumor shrinkage can be maintained in patients with renal cell cancer. Patients will receive ABT-751 by mouth daily for 21 days. Patients will be off drug for 7 days before starting the next cycle of drug.

ELIGIBILITY:
Inclusion Criteria

* Renal Cell Carcinoma.
* Recurrent tumor.
* At least 6 weeks post-nephrectomy.
* Able to tolerate normal activities of daily living.
* Adequate bone marrow, kidney, and liver function.

Exclusion Criteria

* Pregnant or breast feeding.
* Anti-tumor therapy within 4 weeks of the start of ABT-751 administration.
* CNS metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-08; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate in subjects with RCC | 1 year

SECONDARY OUTCOMES:
Time to Tumor Progression (TTP) | 1 year
Survival | 2 years
Toxicities associated with treatment administration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen Eliopoulos, M.D., Study Director — Abbott
Locations (23):
- United States (19):
  - Arizona Cancer Research Center, Tucson, Arizona
  - UCLA School of Medicine, Los Angeles, California
  - Clinical Trials + Research Associates, Montebello, California
  - US Oncology Inc Rocky Mountain Cancer Centers, Denver, Colorado
  - Oncology Hematology Group of South Florida, Miami, Florida
  - US Oncology Inc Florida Cancer Institute, New Port Richey, Florida
  - US Oncology Inc Ocala Oncology Center, Ocala, Florida
  - US Oncology Inc Cancer Centers of Florida, P.A., Orlando, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - US Oncology Inc Raleigh Hematology Oncology Clinic, Cary, North Carolina
  - US Oncology Inc Dayton Oncology & Hematology P.A., Kettering, Ohio
  - US Oncology Inc Cancer Care Accociates-Mercy Campus, Oklahoma City, Oklahoma
  - US Oncology Inc Cancer Centers of the Carolinas, Greenville, South Carolina
  - West Cancer Clinic, Memphis, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - US Oncology Inc Tyler Cancer Center, Tyler, Texas
  - US Oncology Inc Cancer Care Northwest-North, Spokane, Washington
  - US Oncology Inc Northwest Cancer Specialists, Vancouver, Washington
- Canada (4):
  - B.C. Vancouver Cancer Agency, Vancouver, British Columbia
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - McGill University, Montreal, Quebec